CLINICAL TRIAL: NCT05216042
Title: Atrial Natriuretic Peptide and Regulation of Cardiometabolic Health: A Genotype-Guided Human Physiological Study
Brief Title: GENESIS: Genotype Guided - Natriuretic Peptides - Cardiometabolic Health Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Pankaj Arora, MD, Assistant Professor, Division of Cardiovascular Disease, Department of Medicine, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300008758; R01HL163081 (NIH)
Record Dates: First submitted 2022-01-12; First posted 2022-01-31 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases; Natriuretic Peptides; Cardiometabolic Diseases; Energy Expenditure; Glucose Metabolism; Exercise; Obesity
Keywords: Natriuretic Peptides; Cardiovascular Diseases; Glucose Metabolism; Energy Expenditure; Exercise; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Obesity

STUDY DESIGN:
Intervention Model Description: Each participant will be enrolled into one of the two groups based on their genotype.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Low NP Genotype Group (Experimental): 150 healthy adult participants with low NP genotype will be enrolled and each will undergo a physical exam and screening tests to determine participants' eligibility. Participants will consume the study diet for 5 days. On 5th day, the participants will come in for an exercise challenge test. On 6th day, participants will come in a fasting state and drink 75 gm of oral glucose, followed by blood collection every 8 hours.
  Interventions: Dietary Supplement: Study diet; Other: Exercise capacity VO2 max determination; Other: Exercise Challenge; Other: Glucose Challenge
- Active Comparator: High NP Genotype Group (Experimental): 50 healthy adult participants with high NP genotype will be enrolled and each will undergo a physical exam and screening tests to determine participants' eligibility. Participants will consume the study diet for 5 days. On 5th day, the participants will come in for an exercise challenge test. On 6th day, participants will come in a fasting state and drink 75 gm of oral glucose, followed by blood collection every 8 hours.
  Interventions: Dietary Supplement: Study diet; Other: Exercise capacity VO2 max determination; Other: Exercise Challenge; Other: Glucose Challenge

INTERVENTIONS:
Dietary Supplement: Study diet — Participants will consume the study diet for 5 days provided by the clinical research unit's metabolic kitchen (at UAB)
Other: Exercise capacity VO2 max determination — Each participant's maximal oxygen capacity will be determined using a modified Bruce treadmill protocol and will also undergo a DEXA scan to determine the body mass.
Other: Exercise Challenge — Each participant will walk at 70 % of his/her VO2max for 20 minutes on treadmill and will also undergo a resting energy expenditure test.
Other: Glucose Challenge — Participants will come in fasting state on day 6th and will be given 75 gm oral glucose solution to drink, followed by blood collection every hour for next 8 hours.

SUMMARY:
Natriuretic Peptides (NP) are hormones produced by the heart, and they have a wide range of favorable metabolic benefits. Lower levels of these hormones are associated with an increased likelihood of the development of diabetes and poor cardiometabolic health. Obese and Black individuals have ~30% lower levels of NP and are at a greater risk of developing cardiovascular (CV) events as compared to lean and White counterparts. Some people have common genetic variations that cause them to have ~20% lower NP levels. Similar to other low NP populations, these individuals with low NP genotype (i.e., carrying a common genetic variation called rs5068) are at a greater risk of developing cardiometabolic diseases. By understanding the NP response following the exercise challenge and the glucose challenge in individuals with genetically lower NP levels will help us understand how to improve cardiometabolic health in them.

DETAILED DESCRIPTION:
The heart plays an endocrine role by secreting hormones called Natriuretic Peptides (NPs). NPs directly regulates blood pressure (BP) by causing dilation of blood vessels and removing sodium and water from the body. Apart from blood pressure regulation, previous experimental data suggest that NPs has a wide range of favorable metabolic effects and regulates energy homeostasis, fatty acid oxidation, lipid metabolism, glucose intolerance, insulin sensitivity, and obesity. Investigators have demonstrated that low levels of NPs can increase the risk of developing cardiovascular (CV) events (such as heart failure [HF], stroke, myocardial infarction [MI], or heart attack).

Former studies by the investigators have shown that the NP deficient states such as obese and black individuals contributes to lower energy expenditure, poor metabolic profile and promotes the onset of diabetes. Certain genetic factors contribute to the higher predisposition to cardiometabolic disease in individuals with relative atrial natriuretic peptide (ANP) deficiency. PI and others have identified a common genetic variant, rs5068 is associated with higher plasma ANP levels.

The lack of the rs5068 variant has a comparable effect on ANP levels as seen in obese and black individuals and plays a causal role in cardiometabolic health regulation. The rs5068 variant is only present in 10-12% of the population, thereby leaving nearly 90% of adults vulnerable to the potential adverse cardiometabolic impact of having a relative ANP deficiency. This indicates that a low ANP genotype is associated with a poor metabolic health profile.

Our earlier study, in normotensive healthy young adults, demonstrated that a high glucose meal results in reduce ANP levels by 20-30%, which indicates that ANP is a glucose-responsive hormone. The preliminary data from our ongoing clinical trial has shown increased ANP levels with response to the exercise. The impact of genetically determined low ANP levels on the differences in exercise-induced ANP (beneficial) increase and glucose load-induced suppression of ANP (detrimental) is not known in humans.

Micro-RNA-425 (miR-425) is a negative regulator of ANP and acts in a genotype-specific manner. In our previous study, the investigators have demonstrated that miR-425 levels decreased by 71% following one week on a high-salt diet compared with a low-salt diet in individuals with low ANP genotype, and no change was seen in high ANP genotype individuals. In vitro experiments in animals showed an increase in cardiac miR-425 levels by 22-30%. The negative regulator of ANP also independently negatively regulates the control of energy expenditure. The responsiveness of mir-425 to glucose challenge and exercise challenge (metabolic perturbations) has not been previously evaluated in humans.

Individuals with genetically reduced amounts of ANP will be the focus of our present genotype-guided physiological investigation. Following the glucose and exercise challenges, the investigators will additionally investigate the extent to which miR-425 mediated control of ANP suppression occurs. This study will help in understanding how ANP regulates cardiometabolic health in individuals with genetically lower ANP levels.

ELIGIBILITY:
Inclusion Criteria:

* Adults: Age more than or equal to 18; an equal number of Males and Females
* Consent to the collection of genetic material
* Willing to adhere to the study protocol

Exclusion Criteria:

* Age <18, at screening.
* BMI >45 kg/m2.
* Blood pressure more than 140/90 mmHg.
* Participants who are taking more than 2 hypertension medications.
* History of diabetes or fasting plasma glucose >126 mg/dl or HbA1C>=6.5% or prior treatment with antidiabetic medication.
* Have any past or present history of cardiovascular diseases (stroke, seizure, myocardial infarction, heart failure, transient ischemic attack, angina, or cardiac arrhythmia)
* Women who are pregnant or breastfeeding or who can become pregnant and not practicing an acceptable method of birth control during the study (including abstinence);
* Estimated GFR < 60 ml/min/1.73 m2; albumin creatinine ratio ≥30 mg/g
* Hepatic Transaminase (AST and ALT) levels >3x the upper limit of normal
* Anemia (men, Hct < 38%; women, Hct <36%)
* Inability to exercise on a treadmill

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in MRproANP levels following a standardized oral glucose challenge between the high genotype group and low genotype group. | From 1st hour to 8th hour on the main study visit day after consuming study meals for 5 days
Change in Exercise Energy Expenditure between the high genotype and low genotype group. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Change in miR-425 levels following a standardized oral glucose challenge in those with low ANP genotype. | From 1st hour to 8th hour on the main study visit day after consuming study meals for 5 days
Change in miR-425 levels following a standardized exercise challenge in those with low ANP genotype. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days

SECONDARY OUTCOMES:
Change in the NPs (ANP, BNP, NTproBNP) following the glucose challenge between the high genotype group and low genotype group. | From 1st hour to 8th hour on the main study visit day after consuming study meals for 5 days
Change in the serum glucose following the glucose challenge between the high genotype group and low genotype group. | From 1st hour to 8th hour on the main study visit day after consuming study meals for 5 days
Change in the serum insulin following the glucose challenge between the high genotype group and low genotype group. | From 1st hour to 8th hour on the main study visit day after consuming study meals for 5 days
Change in Resting Energy Expenditure (REE) between the two genotype groups. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Change in the NPs (ANP, BNP, NTproBNP) with standardized exercise protocol between the two genotype groups. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Change in the serum glucose levels with standardized exercise protocol between the two genotype groups. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Change in the serum insulin levels with standardized exercise protocol between the two genotype groups. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Change in the free fatty acid levels with standardized exercise protocol between the two genotype groups. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Change in the glycerol levels with standardized exercise protocol between the two genotype groups. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Change in miR-425 levels with change in NP levels (ANP, MRproANP, BNP, and NTproBNP) following glucose challenge. | From 1st hour to 8th hour on the main study visit day after consuming study meals for 5 days
Change in miR-425 levels with change in NP levels (ANP, MRproANP, BNP, and NTproBNP) following exercise challenge. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Change in miR-425 levels with change in serum glucose levels following glucose challenge. | From 1st hour to 8th hour on the main study visit day after consuming study meals for 5 days
Change in miR-425 levels with change in serum insulin levels following glucose challenge. | From 1st hour to 8th hour on the main study visit day after consuming study meals for 5 days
Change in miR-425 levels with change in serum glucose levels following exercise challenge. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Change in miR-425 levels with change in serum insulin levels following exercise challenge. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Correlation of resting miR-425 levels with REE | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
  Levels of miR-425 measured in 2-ΔΔCT will be assessed and will be related to REE measured in kcal/min
Change in miR-425 levels with change in NP levels (ANP, MRproANP, BNP, and NTproBNP) following glucose challenge between the two genotype groups. | From 1st hour to 8th hour on the main study visit day after consuming study meals for 5 days
Change in miR-425 levels with change in NP levels (ANP, MRproANP, BNP, and NTproBNP) following exercise challenge between the two genotype groups. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Change in miR-425 levels with change in serum glucose levels following glucose challenge between the two genotype groups. | From 1st hour to 8th hour on the main study visit day after consuming study meals for 5 days
Change in miR-425 levels with change in serum insulin levels following glucose challenge between the two genotype groups. | From 1st hour to 8th hour on the main study visit day after consuming study meals for 5 days
Change in miR-425 levels with change in serum glucose levels following exercise challenge between the two genotype groups. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Change in miR-425 levels with change in serum insulin levels following exercise challenge between the two genotype groups. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
Correlation of resting miR-425 levels with REE between the genotype groups. | About 3 hours on the exercise challenge visit day after consuming study meals for 4 days
  Levels of miR-425 levels measured in 2-ΔΔCT will be related to the REE measured in kcal/min and will be compared between the genotype groups

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Arora, MD, FAHA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parcha V, Patel N, Gutierrez OM, Li P, Gamble KL, Musunuru K, Margulies KB, Cappola TP, Wang TJ, Arora G, Arora P. Chronobiology of Natriuretic Peptides and Blood Pressure in Lean and Obese Individuals. J Am Coll Cardiol. 2021 May 11;77(18):2291-2303. doi: 10.1016/j.jacc.2021.03.291. PMID 33958126
- [Background] Arora P, Wu C, Hamid T, Arora G, Agha O, Allen K, Tainsh RET, Hu D, Ryan RA, Domian IJ, Buys ES, Bloch DB, Prabhu SD, Bloch KD, Newton-Cheh C, Wang TJ. Acute Metabolic Influences on the Natriuretic Peptide System in Humans. J Am Coll Cardiol. 2016 Feb 23;67(7):804-812. doi: 10.1016/j.jacc.2015.11.049. PMID 26892417
- [Background] Bajaj NS, Gutierrez OM, Arora G, Judd SE, Patel N, Bennett A, Prabhu SD, Howard G, Howard VJ, Cushman M, Arora P. Racial Differences in Plasma Levels of N-Terminal Pro-B-Type Natriuretic Peptide and Outcomes: The Reasons for Geographic and Racial Differences in Stroke (REGARDS) Study. JAMA Cardiol. 2018 Jan 1;3(1):11-17. doi: 10.1001/jamacardio.2017.4207. PMID 29167879
- [Background] Arora P, Reingold J, Baggish A, Guanaga DP, Wu C, Ghorbani A, Song Y, Chen-Tournaux A, Khan AM, Tainsh LT, Buys ES, Williams JS, Heublein DM, Burnett JC, Semigran MJ, Bloch KD, Scherrer-Crosbie M, Newton-Cheh C, Kaplan LM, Wang TJ. Weight loss, saline loading, and the natriuretic peptide system. J Am Heart Assoc. 2015 Jan 16;4(1):e001265. doi: 10.1161/JAHA.114.001265. PMID 25595796
- [Background] Parcha V, Kalra R, Li P, Oparil S, Arora G, Arora P. Nocturnal blood pressure dipping in treated hypertensives: insights from the SPRINT trial. Eur J Prev Cardiol. 2022 Feb 19;29(1):e25-e28. doi: 10.1093/eurjpc/zwaa125. No abstract available. PMID 33624057